CLINICAL TRIAL: NCT01284933
Title: Carotid Plaque Imaging in Acute Stroke
Acronym: CAPIAS
Status: Completed | Type: Observational
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Martin Dichgans, Prof., Ludwig-Maximilians - University of Munich
Other Study IDs: ISD-CAPIAS-01
Record Dates: First submitted 2011-01-24; First posted 2011-01-27 (Estimated); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Stroke; Ischemic Attack, Transient
Keywords: Stroke; Ischemic Attack, Transient; Magnetic Resonance Imaging; Carotid Arteries; Carotid Artery Plaque; Atherosclerosis
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient; Carotid Stenosis; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, plasma, RNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute Ischemic Stroke, TIA: Patients admitted to a specialized stroke service because of an acute ischemic stroke or a transient ischemic attack (TIA).

SUMMARY:
The purpose of this study is to determine the frequency, characteristics, and consequences of vulnerable carotid artery plaques ipsilateral to an acute ischemic stroke or TIA in the territory of the internal carotid artery.

DETAILED DESCRIPTION:
Even with extensive diagnostic workup the underlying etiology remains unidentified in about 25% of patients with acute ischemic stroke (AIS) or transient ischemic attack (TIA). Non-invasive high-resolution magnetic resonance imaging (HR-MRI) of the carotid artery allows detecting vulnerable plaques (VP) and quantifying single plaque components. The hypotheses behind this study are that i) a substantial proportion of cases of AIS and TIA within the anterior circulation and no identified cause (cryptogenic AIS or TIA) are caused by VP in the carotid artery; ii) that these patients are at a high risk of developing a recurrent stroke, TIA, or clinically silent lesions detectable by brain MRI; and iii) that VP in the carotid artery are associated with specific infarct patterns as detected by diffusion-weighted MR imaging. Finally, the investigators will search for biomarkers associated with vulnerable carotid artery plaques. Motivating this study are the following considerations: i) data on the frequency and characteristics of VP in patients with cryptogenic AIS or TIA will provide valuable insights into stroke mechanisms; ii) depending on the results this study may have implications for diagnostic decision making and provide the basis for the planning of targeted interventional studies.

ELIGIBILITY:
Inclusion Criteria:

* Age > 49 years old
* Acute ischemic stroke or transient ischemic attack (TIA)
* Neurological symptoms compatible with a stroke or TIA in the anterior circulation (territory of the internal carotid artery)
* Onset of symptoms within the last 7 days
* 1 or more acute ischemic lesion(s) visible on MR diffusion-weighted imaging (DWI) in the territory of a single internal carotid artery
* Presence of carotid artery plaques in the ipsilateral or contralateral carotid artery as defined by ultrasound (criteria: plaque thickness at least 2mm; located within 1cm proximal or distal to the carotid bifurcation)
* Written informed consent

Exclusion Criteria:

* Primary referral to an outside hospital (to avoid recruitment bias)
* DWI positive lesions outside the territory of a single internal carotid artery
* Carotid artery stenosis > 69% (North American Symptomatic Carotid Endarterectomy Trial (NASCET) criteria) ipsilateral to the stroke or TIA as defined by ultrasound (systolic peak flow velocity ≥ 300 cm/s)
* Standard contra-indications for MRI
* Documented allergy to MRI contrast media
* History of radiation to the neck area
* Renal clearance < 30 ml/minute
* Creatinine levels > 2 times the upper limit of the standard range of the respective laboratory within the last 30 days prior to MRI
* Surgical procedure within 24 hours preceding the MRI

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to a specialized stroke service because of an acute stroke or TIA
Sampling Method: Probability Sample
Enrollment: 234 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2021-07 (Actual)

PRIMARY OUTCOMES:
Frequency and characteristics of vulnerable plaques (VP) in the carotid artery ipsilateral to an acute ischemic stroke (AIS) or TIA in the territory of the carotid artery in patients with a cryptogenic stroke | Baseline
  For the primary outcome, definition of a VP will be based on non-invasive high-resolution magnetic resonance imaging (MRI). We will classify plaques according to the American Heart Association - Lesion Type (AHA-LT) classification (Cai et al. Circulation 2002; Saam et al.).
  Comparisons will include:
  * a comparison of the frequency and characteristics of VP ipsilateral vs. contralateral to the AIS or TIA
  * a comparison of the frequency and characteristics of ipsilateral VP in patients with cryptogenic stroke as compared to patients with cardioembolic stroke or small vessel stroke

SECONDARY OUTCOMES:
Pattern of acute ischemic lesions on brain MRI associated with VP in the carotid artery | Baseline
  The pattern of acute ischemic lesions on brain MRI associated with VP in the carotid artery will be analyzed.
Recurrence rates of AIS or TIA in patients with VP in the carotid artery | 12, 24, 36 Months
  The recurrence rates of acute ischemic strokes or transient ischemic attacks will be evaluated at follow-up after 12, 24 and 36 months.
Rate of new ischemic lesions on FLAIR MRI at 12 month follow-up in patients with VP in the carotid artery | 12 Months
  The rate of new ischemic lesions on FLAIR MRI will be evaluated at follow-up after 12 months.
Association between VP in the carotid artery and atherosclerotic plaques in the aortic arch as determined by transoesophageal ultrasound | Baseline
  The association between VP in the carotid artery and atherosclerotic plaques in the aortic arch as determined by transoesophageal ultrasound will be evaluated in patients with transoesophageal ultrasound.
Biomarkers associated with vulnerable carotid artery plaques | Baseline
  Biomarkers probably associated with vulnerable carotid artery plaques will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Dichgans, Prof., Principal Investigator — Institute for Stroke and Dementia Research, Klinikum der Universität München; Tobias Saam, Prof., Principal Investigator — Department of Radiology, Klinikum der Universität München
Locations (4):
- Germany (4):
  - University of Freiburg, Germany, Freiburg im Breisgau, Baden-Wurttemberg
  - Interdisciplinary Stroke Center Munich, Klinikum der Universität München, Munich, Bavaria
  - Klinikum re. der Isar, Technical University Munich, Munich, Bavaria
  - University of Tuebingen, Tübingen

REFERENCES:
- [Background] Bayer-Karpinska A, Schwarz F, Wollenweber FA, Poppert H, Boeckh-Behrens T, Becker A, Clevert DA, Nikolaou K, Opherk C, Dichgans M, Saam T. The carotid plaque imaging in acute stroke (CAPIAS) study: protocol and initial baseline data. BMC Neurol. 2013 Dec 13;13:201. doi: 10.1186/1471-2377-13-201. PMID 24330333
- [Background] Schwarz F, Bayer-Karpinska A, Poppert H, Buchholz M, Cyran C, Grimm J, Helck A, Nikolaou K, Opherk C, Dichgans M, Saam T. Serial carotid MRI identifies rupture of a vulnerable plaque resulting in amaurosis fugax. Neurology. 2013 Mar 19;80(12):1171-2. doi: 10.1212/WNL.0b013e31828869ad. No abstract available. PMID 23509049
- [Result] Kopczak A, Schindler A, Bayer-Karpinska A, Koch ML, Sepp D, Zeller J, Strecker C, Hempel JM, Yuan C, Malik R, Wollenweber FA, Boeckh-Behrens T, Cyran CC, Helck A, Harloff A, Ziemann U, Poli S, Poppert H, Dichgans M, Saam T. Complicated Carotid Artery Plaques as a Cause of Cryptogenic Stroke. J Am Coll Cardiol. 2020 Nov 10;76(19):2212-2222. doi: 10.1016/j.jacc.2020.09.532. PMID 33153580
- [Derived] Kopczak A, Schindler A, Sepp D, Bayer-Karpinska A, Malik R, Koch ML, Zeller J, Strecker C, Janowitz D, Wollenweber FA, Hempel JM, Boeckh-Behrens T, Cyran CC, Helck A, Harloff A, Ziemann U, Poli S, Poppert H, Saam T, Dichgans M. Complicated Carotid Artery Plaques and Risk of Recurrent Ischemic Stroke or TIA. J Am Coll Cardiol. 2022 Jun 7;79(22):2189-2199. doi: 10.1016/j.jacc.2022.03.376. Epub 2022 May 3. PMID 35523659
- [Derived] Kopczak A, Schindler A, Dichgans M, Saam T. Reply: Comparison of Different Plaque Imaging Techniques to Detect Complicated Carotid Artery Plaques. J Am Coll Cardiol. 2021 Mar 2;77(8):1147-1148. doi: 10.1016/j.jacc.2020.12.038. No abstract available. PMID 33632492
- See also: Click here for more information — http://www.klinikum.uni-muenchen.de/Interdisziplinaeres-Schlaganfallzentrum/en/index.html
- See also: Click here for more information — http://www.klinikum.uni-muenchen.de/Institut-fuer-Schlaganfall-und-Demenzforschung/en/index.html